CLINICAL TRIAL: NCT02646735
Title: A Randomized, Open Label, Multi-Centre Study to Compare the Efficacy and Tolerability of Fulvestrant 500mg With Exemestane for Postmenopausal Advanced Breast Cancer Patients
Brief Title: Fulvestrant 500mg With Exemestane Endocrine Therapy for Postmenopausal Advanced Breast Cancer Patients
Acronym: FRIEND
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Binghe Xu, Head of the medical department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10982
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fulvestrant (Experimental): Fulvestrant 500 mg
  Interventions: Drug: Fulvestrant 500 mg
- Exemestane (Active Comparator): Exemestane 25mg
  Interventions: Drug: Exemestane 25 mg

INTERVENTIONS:
Drug: Fulvestrant 500 mg — Fulvestrant 500mg will be given monthly.
  Arms: Fulvestrant
Drug: Exemestane 25 mg — Exemestane 25mg will be given once daily.
  Arms: Exemestane

SUMMARY:
A Randomized, Open label, Parallel-group, Multi-center study. Eligible patients will be randomized in a 1:1 ratio to receive fulvestrant 500 mg or Exemestane 25mg.

DETAILED DESCRIPTION:
To compare the efficacy and tolerability of Fulvestrant 500 mg with Exemestane 25 mg as first line endocrine therapy in postmenopausal women with oestrogen receptor positive HER2 negative advanced breast cancer who have relapsed on or after adjuvant non-aromatase inhibitor therapy

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent document on file;
* Age over 60 years;
* Age < 60 years and amenorrheic for 12 or more months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression and FSH and oestradiol level in the postmenopausal range;
* Patients with metastatic or locally advanced disease not amenable to therapy with Curative intent
* ER + and/or PgR +;
* Duration of adjuvant non-aromatase inhibitors treatment should be at least 2 years or more;
* WHO performance status 0, 1 or 2;
* Patients with life expectancy of more than 3 months.

Exclusion Criteria:

* Presence of life-threatening metastatic visceral disease;
* Previous systemic chemotherapy for advanced breast cancer;
* Received systemic endocrine therapy for advanced disease;
* Extensive radiation therapy within the last 4 weeks ;
* Platelets < 100*109 / L,Total bilirubin no less than 1.5ULRR, ALT or AST no less than 2.5ULRR if no demonstrable liver metastases or no less than 5ULRR in presence of liver metastases;
* Severe renal impairment, bleeding diathesis, long-term anticoagulant therapy;
* History of hypersensitivity to active or inactive excipients of fulvestrant, Exemestane and/or castor oil.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
PFS | 3 years
  To compare the efficacy of Fulvestrant 500 mg with the patients treated with Exemestane 25mg as first line setting in terms of progression-free survival.

SECONDARY OUTCOMES:
ORR | 3 years
  To compare the objective response rate of patients treated with Fulvestrant 500 mg with Exemestane.

CONTACTS AND LOCATIONS:
Overall Officials: XU Binghe, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Institute, Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Cai L, Song Y, Sun T, Tong Z, Teng Y, Li H, Ouyang Q, Chen Q, Cui S, Yin Y, Liao N, Sun Q, Feng J, Wang X, Xu B. Clinical efficacy of fulvestrant versus exemestane as first-line therapies for Chinese postmenopausal oestrogen-receptor positive /human epidermal growth factor receptor 2 -advanced breast cancer (FRIEND study). Eur J Cancer. 2023 May;184:73-82. doi: 10.1016/j.ejca.2023.02.007. Epub 2023 Feb 15. PMID 36905771